CLINICAL TRIAL: NCT05531045
Title: 18F-FDG Positron Emission Tomography/Tomodensitometry for Early Evaluation of Chemotherapy Efficacy in Metastatic Colic Adenocarcinoma
Brief Title: 18FFDG PET/CT for Early Evaluation of Chemotherapy Efficacy in Metastatic Colic Adenocarcinoma
Acronym: TEP-PREDICT
Status: Not yet recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP180576
Record Dates: First submitted 2022-08-11; First posted 2022-09-07 (Actual); Last update posted 2022-09-07 (Actual); Status verified 2022-08

CONDITIONS: Metastatic Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Positron Emission Tomography Computed Tomography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cohort: FDG PET/CT assessed after 2 cycles of chemotherapy
  Interventions: Diagnostic Test: PET/CT

INTERVENTIONS:
Diagnostic Test: PET/CT — FDG PET/CT assessed after 2 cycles of chemotherapy with PERCIST criteria

SUMMARY:
The metastatic colo-rectal cancer (especially with hepatic metastatic lesions, but also peritoneal or pulmonary lesions) is a major public health issue, because of its frequency, the heavy treatments and the cost of new therapeutic molecules involved, in particular targeted therapies that can result in specific adverse events. The first-line treatment often consists of a polychemotherapy, which can be associated to a targeted therapy. According to the therapeutic response, patient condition and disease extent, some patients may benefit from prognosis-changing treatments such as surgery of metastases. However, the best morphological response is most of time evidenced after only 6 or 8 cycles of treatment, corresponding to 3 to 4 months. Therapeutic evaluation with FDG PET/CT is validated in several neoplasia (lymphoma, breast cancer). Data on FDG PET evaluation of colic cancer chemotherapy are currently insufficient to propose its use in the usual clinical setting. We thus are going to study the performance of early FDG PET therapeutic evaluation to predict response to first-line chemotherapy in patients with potentially resectable metastases. If early PET diagnostic performances prove satisfying, this approach could become of paramount importance to tailor therapeutic strategy for these patients, with the possibility of early modification of chemotherapy protocol, which is now possible thanks to the existence of therapeutic alternatives (chemotherapy intensification, replacement of oxaliptaine by irinotecan or conversely, replacement of an anti-EGFR by an anti-angiogenic or conversely).

ELIGIBILITY:
Inclusion Criteria:

* Histologically proved colo-rectal cancer
* Measurable metastatic disease according to RECIST 1.1 criteria
* Metastases considered potentially resectable (for example : hepatic, nodular peritoneal, lung lesions…) by the multidisciplinary committee meeting
* ECOG≤2
* Patient candidate to a first-line chemotherapy± targeted therapy according to standard protocols : LV5FU2, FOLFOX, FOLFIRI, FOLFIRINOX +/- bévacizumab, aflibercept , cétuximab, panitumumab
* In case of metachrone metastasis, adjuvant chemotherapy stopped for more than 6 months before relapse diagnosis
* Predictable life expectancy of more than 6 months
* Signed informed consent
* Age > 18 years

Exclusion Criteria:

* Patient with another evolutive neoplastic disease
* Patient participating in another study evaluating an imaging technique using ionizing radiations
* Brain metastasis
* Absence of health insurance coverage
* Pregnant of breastfeeding woman
* Hypersensitivity to FDG or to one of the excipients of used specialty

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Population fo patients with metastic colo-rectal cancer eligible to first line chemotherapy
Sampling Method: Non-Probability Sample
Enrollment: 222 (Estimated)
Dates: Start 2022-09 (Estimated); Primary Completion 2025-01 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
early metabolic response assessed by PERCIST criteria | 4 months

SECONDARY OUTCOMES:
Resection of metastases defined by a R0 or R1 resection (macroscopically complete surgery with disease-free margins or minimal residual disease) after the end of first line chemotherapy | at the end of first line chemotherapy, an average of 12 months
Best morphological response during the course of first line chemotherapy | at the end of first line chemotherapy, an average of 12 months
percentage of cases where early metabolic response evaluation would have led to a modification of the therapeutic strategy/management | Month 2
Progression Free Survival | 36 months
Overall Survival | 36 months
ΔSUVmax (EORTC criteria) between Pre-therapeutic and 2 cycles PET assessment | 2 months
ΔSULpeak (PERCIST criteria) between Pre-therapeutic and 2 cycles PET assessment | 2 months
ΔMTV between Pre-therapeutic and 2 cycles PET assessment | 2 months
ΔTLG between Pre-therapeutic and 2 cycles PET assessment | 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Aparicio, MD, Study Director — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital Saint Louis, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided